CLINICAL TRIAL: NCT03339284
Title: Quadratus Lumborum Block (QLB) With and Without Dexamethasone: the Effect on Postoperative Pain and Recovery After Laparoscopic Nephrectomy
Brief Title: QLB and Laparoscopic Nephrectomy, Postoperative Pain and Recovery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R17103M; 2017-002254-37 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Pain; Chronic Pain Post-Proceduraal; Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — dexamethasone 21-phosphate; Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are randomized and allocated in blocks of nine to either placebo or QLB with dexamethasone or QLB without dexamethasone group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QLB with dexamethasone (Active Comparator): Single sided US-guided QLB using ropivacaine 3,75 mg/ml 20 ml and dexamethasone 5 mg/ml 0,4 ml
  Interventions: Drug: Dexamethasone sodium phosphate; Drug: Ropivacaine Hydrocloride
- QLB without dexamethasone (Active Comparator): Single sided US-guided QLB using ropivacaine 3,75 mg/ml 20 ml and isotonic natriumchloride solution (NaCl 0,9%) 0,4 ml
  Interventions: Drug: Ropivacaine Hydrocloride; Drug: Sodium Chloride 9mg/mL
- Placebo (Placebo Comparator): Single sided US-guided QLB using isotonic natriumchloride solution (NaCl 0,9%) 20,4 ml
  Interventions: Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — Dexamethasone injection
  Other Names: Oradexon
  Arms: QLB with dexamethasone
Drug: Ropivacaine Hydrocloride — Ropivacaine injection
  Arms: QLB with dexamethasone; QLB without dexamethasone
Drug: Sodium Chloride 9mg/mL — Sodium Chloride injection
  Other Names: Saline
  Arms: Placebo; QLB without dexamethasone

SUMMARY:
There are ca 900 new cases of kidney cancer in Finland/year. The curative therapy for kidney cancer is partial or total nephrectomy depending on the localization and the size of tumor. Main of these operations are laparoscopic.

Epidural analgesia is considered as most effective for the treatment of postoperative pain after open nephrectomy, but after laparoscopic operation parenteral and enteral opioids combined with paracetamol (acetaminophen) usually offer adequate postoperative pain relief. However, the need for opioids postoperatively may be high and side effects, such as sedation and nausea, are common. On the other hand epidural analgesia has some contraindications and risks for serious complications. Nevertheless, inadequately treated acute postoperative pain is considered as one of the main risk factors for persistent postoperative pain.

Recently quadratus lumborum block (QLB) has gained popularity in the treatment of postoperative pain after various surgeries in the area from hip to mamilla. It is more beneficial than other peripheral blocks, since it covers also the visceral nerves. A single shot QLB has reported to last up to 48 hours.

Perineural dexamethasone added to local anesthetic has been reported to prolong the duration of analgesia of the perineural nerve block, but it's effect on the duration of QLB is not known.

90 kidney cancer patients with planned laparoscopic nephrectomy aging 18-85 will be recruited based on a power calculation. The primary outcome measure is the postoperative cumulative opioid consumption. Secondary outcomes are acute pain (NRS scale), nausea, vomiting, mobilisation and long term outcomes such as quality of life and persistent pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with renal cancer coming to the laparoscopic radical nephrectomy

Exclusion Criteria:

* age under 18y or over 85y
* diabetes type 1 with complications
* no co-operation or inadequate finnish language skills
* persistent pain for other reason
* severe hepatic insufficiency or paracetamol (acetaminophen) is contraindicated for other reason
* any type of steroid in regular use
* oxycodone contraindicated
* medications changing notably paracetamol (acetaminophen) and/or ropivacaine metabolism in regular use

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
opiate consumption | 24 hours
  cumulative opiate consumption postoperatively

SECONDARY OUTCOMES:
opiate consumption | 72 hours
  cumulative opiate consumption postoperatively
postoperative nausea | 72 hours
  numerical rating scale
pain score | 7 days
  numerical rating scale
mobilization | 72 hours
  time to standing up and mobilizing after surgery
quality of life | 12 months
  SF36 query
persistent pain | 12 months
  paindetect McGill
functional query | 12 months
  assessment how pain in operation region limits daily functions
postoperative vomiting | 72 hours
  amount of vomites

CONTACTS AND LOCATIONS:
Overall Officials: Maija Kalliomaki, PhD, Principal Investigator — Tampere University Hospital, Department of Anesthesia
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finnish Cancer Registry. Cancer in Finland 2007-2011. Cancer Society of Finland Publication, Helsinki.
- [Background] Ljungberg B, Bensalah K, Canfield S, Dabestani S, Hofmann F, Hora M, Kuczyk MA, Lam T, Marconi L, Merseburger AS, Mulders P, Powles T, Staehler M, Volpe A, Bex A. EAU guidelines on renal cell carcinoma: 2014 update. Eur Urol. 2015 May;67(5):913-24. doi: 10.1016/j.eururo.2015.01.005. Epub 2015 Jan 21. PMID 25616710
- [Background] Chan DY, Cadeddu JA, Jarrett TW, Marshall FF, Kavoussi LR. Laparoscopic radical nephrectomy: cancer control for renal cell carcinoma. J Urol. 2001 Dec;166(6):2095-9; discussion 2099-100. doi: 10.1016/s0022-5347(05)65513-9. PMID 11696714
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956
- [Background] Kirksey MA, Haskins SC, Cheng J, Liu SS. Local Anesthetic Peripheral Nerve Block Adjuvants for Prolongation of Analgesia: A Systematic Qualitative Review. PLoS One. 2015 Sep 10;10(9):e0137312. doi: 10.1371/journal.pone.0137312. eCollection 2015. PMID 26355598
- [Background] Huynh TM, Marret E, Bonnet F. Combination of dexamethasone and local anaesthetic solution in peripheral nerve blocks: A meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2015 Nov;32(11):751-8. doi: 10.1097/EJA.0000000000000248. PMID 25774458
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Gordon DB, de Leon-Casasola OA, Wu CL, Sluka KA, Brennan TJ, Chou R. Research Gaps in Practice Guidelines for Acute Postoperative Pain Management in Adults: Findings From a Review of the Evidence for an American Pain Society Clinical Practice Guideline. J Pain. 2016 Feb;17(2):158-66. doi: 10.1016/j.jpain.2015.10.023. Epub 2015 Dec 21. PMID 26719073
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Gustavsson A, Bjorkman J, Ljungcrantz C, Rhodin A, Rivano-Fischer M, Sjolund KF, Mannheimer C. Socio-economic burden of patients with a diagnosis related to chronic pain--register data of 840,000 Swedish patients. Eur J Pain. 2012 Feb;16(2):289-99. doi: 10.1016/j.ejpain.2011.07.006. PMID 22323381
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500